CLINICAL TRIAL: NCT03386214
Title: Pevonedistat in Combination With Ruxolitinib for Treatment of Patients With Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor stopped development of pevonedistat
Sponsor: Washington University School of Medicine (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201802152; IISR-2017-101916 (Other: Takeda)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Myelofibroses
MeSH Terms: conditions — Primary Myelofibrosis | interventions — pevonedistat; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Starting Dose - 5 mg/m^2 pevonedistat + ruxolitinib (Experimental): * Pevonedistat will be given as an IV infusion at the assigned dose over the course of 60 minutes on Days 1, 3, and 5 of each 28-day cycle.
  * Ruxolitinib will be continued at the same dose as prior to enrollment and will be administered as standard of care outside the study protocol.
  Interventions: Drug: Pevonedistat; Drug: Ruxolitinib; Procedure: Peripheral blood draw; Procedure: Skin biopsy
- Arm 2: Dose Level 2 - 10 mg/m^2 pevonedistat + ruxolitinib (Experimental): * Pevonedistat will be given as an IV infusion at the assigned dose over the course of 60 minutes on Days 1, 3, and 5 of each 28-day cycle.
  * Ruxolitinib will be continued at the same dose as prior to enrollment and will be administered as standard of care outside the study protocol.
  Interventions: Drug: Pevonedistat; Drug: Ruxolitinib; Procedure: Peripheral blood draw; Procedure: Skin biopsy
- Arm 3: Dose Level 3 - 20 mg/m^2 pevonedistat + ruxolitinib (Experimental): * Pevonedistat will be given as an IV infusion at the assigned dose over the course of 60 minutes on Days 1, 3, and 5 of each 28-day cycle.
  * Ruxolitinib will be continued at the same dose as prior to enrollment and will be administered as standard of care outside the study protocol.
  Interventions: Drug: Pevonedistat; Drug: Ruxolitinib; Procedure: Peripheral blood draw; Procedure: Skin biopsy

INTERVENTIONS:
Drug: Pevonedistat — The amount of pevonedistat to be administered will be based on body surface area (BSA). BSA will be calculated using a standard formula on Cycle 1 Day 1, and on Day 1 of subsequent cycles if the patient experiences a > 5% change in body weight from the weight used for the most recent BSA calculation.
  Other Names: MLN4924
Drug: Ruxolitinib — -Standard of care outside of protocol
  Other Names: Jakavi®
Procedure: Peripheral blood draw — * Baseline or Cycle 1 Day 1 (prior to study treatment administration)
  * Cycle 2 Day 1 (prior to study treatment administration)
  * Cycle 4 Day 1 (prior to study treatment administration)
  * End of treatment
Procedure: Skin biopsy — A skin punch biopsy specimen will be collected at the baseline visit. One 6 mm punch biopsy of normal skin will be performed using standard techniques and local anesthesia.

SUMMARY:
Based on the investigators' preclinical data, the combination of pevonedistat and ruxolitinib may provide greater clinical responses in patients with myelofibrosis compared to ruxolitinib monotherapy via inhibition of NFκB in addition to JAK-STAT signaling.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary myelofibrosis or post-polycythemia vera/essential thrombocythemia myelofibrosis classified as high risk, intermediate-2 risk, or intermediate 1 risk by IPSS.
* On treatment with ruxolitinib for at least 3 months and have been on a stable dose for at least 8 weeks and have not achieved a CR by IWG criteria.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 500/mcL, and have not received any growth factor support for at least 4 weeks prior to screening
  * Platelets ≥ 50,000/mcL
  * Peripheral blood blasts ≤ 10%
  * Albumin > 2.7 g/dL
  * Total bilirubin ≤ institutional upper limit of normal (IULN); patients with Gilbert's syndrome may enroll if direct bilirubin ≤ 1.5 x IULN
  * ALT and AST ≤ 2.5 x IULN
  * Creatinine clearance ≥ 50 mL/min
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential:

    * Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, status postvasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* History of allogeneic stem cell transplant.
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during the study period.
* Received hydroxyurea therapy within 28 days (4 weeks) before the first dose of any study drug.
* Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 14 days before the first dose of any study drug.
* Currently receiving any other investigational agents.
* Treatment with clinically significant metabolic enzyme inducers within 14 days before the first dose of study drug. Clinically significant metabolic enzyme inducers are not permitted during the study.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pevonedistat, ruxolitinib, or other agents used in the study.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.
* Diagnosis or treated for another malignancy within 2 years before enrollment, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any time are not excluded if they have undergone resection.
* Ongoing or active infection.
* Known cardiopulmonary disease defined as:

  * Unstable angina pectoris
  * Congestive heart failure (NYHA class III or IV)
  * Myocardial infarction within 6 months prior to first dose (patients who had ischemic heart disease such as ACS, MI, and/or revascularization more than 6 months prior to enrollment and who are without cardiac symptoms may enroll)
  * Symptomatic cardiomyopathy
  * Clinically significant cardiac arrhythmia

    * History of polymorphic ventricular fibrillation or Torsade de Pointes
    * Permanent atrial fibrillation (a fib), defined as continuous a fib for ≥ 6 months
    * Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening
    * Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g. pacemaker) or ablation. Patients with Paroxysmal a fib or < grade 3 a fib for a period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen.
    * Implantable cardioverter defibrillator
    * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing)
* Clinically significant pulmonary hypertension requiring pharmacologic therapy
* Uncontrolled coagulopathy or bleeding disorder.
* Uncontrolled high blood pressure (i.e. systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg).
* Prolonged rate corrected QT (QTc) interval ≥ 500 msec, calculated according to institutional guidelines.
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography.
* Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, or pulmonary fibrosis.
* Known hepatic cirrhosis or severe pre-existing hepatic impairment.
* Known CNS involvement.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Female patients who intend to donate eggs and male patients who intended to donate sperm during the course of this study or for 4 months after receiving the last dose of study treatment.
* Female patients who are both lactating and breastfeeding or have positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug
* Known HIV-positivity.
* Chronic, active, or acute viral hepatitis A, B, or C infection, or hepatitis B or C carrier.
* Life-threatening illness unrelated to cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of pevonedistat in combination with ruxolitinib in patients with myelofibrosis as measured by the frequency of adverse events | Through 30 days after completion of treatment (estimated to be 42 weeks)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Safety and tolerability of pevonedistat in combination with ruxolitinib in patients with myelofibrosis as measured by the maximum tolerated dose (MTD) | 28 days after enrollment of last participant (estimated to be 25 months)
  -MTD: The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached.

SECONDARY OUTCOMES:
Spleen response with the combination of pevonedistat and ruxolitinib | Through 12 weeks after completion of treatment (estimated to be 48 weeks)
  * A baseline splenomegaly that is palpable at 5-10 cm below the left costal margin becomes not palpable OR
  * A baseline splenomegaly that is palpable > 10 cm below the left costal margin decreases by ≥50% OR
  * A baseline splenomegaly that is palpable < 5 cm below the left costal margin is not eligible for spleen response OR
  * Ultrasound shows ≥35% spleen volume reduction (calculated)
Improvement of constitutional symptoms with the combination of pevonedistat and ruxolitinib | Through completion of treatment (estimated to be 36 weeks)
  * A ≥50% reduction in the myeloproliferative neoplasm symptom assessment total symptom score
  * 8 symptoms (tiredness, early satiety, abdominal discomfort, inactivity, night sweats, itching, bone pain, pain under ribs under left side) with 0 to 10 ranking where 0=no pain and 10=worst imaginable pain
Hematologic response with the combination of pevonedistat and ruxolitinib as measured by anemia response | Through 12 weeks after completion of treatment (estimated to be 48 weeks)
  -Anemia response is only applicable for patients with a baseline hemoglobin level less than 10g/dL for 8 weeks or more, and requires:
  * ≥ 2 g/dL increase in hemoglobin level OR
  * becoming transfusion-independent (no RBC transfusions in past 1 month)
Hematologic response with the combination of pevonedistat and ruxolitinib as measured by platelet response | Through 12 weeks after completion of treatment (estimated to be 48 weeks)
  -Platelet response is only applicable for patients with a baseline platelet count of less than 50 x 109/L for 8 weeks or more, and requires:
  * 100% increase in platelet count AND
  * An absolute platelet count of at least 50 x 109/L
Pharmacokinetics of pevonedistat when co-administered with ruxolitinib as measured by the Cmax (peak serum concentration) | Through Cycle 1 Day 5
Pharmacokinetics of pevonedistat when co-administered with ruxolitinib as measured by the Tmax (time of maximum concentration observed) | Through Cycle 1 Day 5
Pharmacokinetics of pevonedistat when co-administered with ruxolitinib as measured by the area under the plasma drug concentration curve (AUC) | At 24 hours
  -AUC reflects the actual body exposure to drug after administration of a dose of the drug and is expressed

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Oh, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu